CLINICAL TRIAL: NCT04892849
Title: Clinical Benefit and Biomarker Analysis of Combination of PD-1/PD-L1 Immune Checkpoint Inhibitors and Radiotherapy in NSCLC, HNSCC and Other Solid Tumors
Brief Title: Clinical Benefit and Biomarker Analysis of Combination of PD-1/PD-L1 Immune Checkpoint Inhibitors and Radiotherapy
Acronym: ST-ICI02
Status: Recruiting | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: ST-ICI02
Record Dates: First submitted 2021-04-26; First posted 2021-05-19 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: HNSCC; NSCLC; Esophageal Cancer; Urothelial Carcinoma; Renal Cell Carcinoma; Squamous Cell Carcinoma of the Skin; Small Cell Bronchial Carcinomas
Keywords: Immunotherapy; Radiotherapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Esophageal Neoplasms; Carcinoma, Transitional Cell; Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, serum, plasma, immunecell RNA, immunecell DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Trial cohort: The study cohort consist of patients suffering from HNSCC (palliative), NSCLC (separately palliative and adjuvant) and "other solid tumors" (including in particular esophageal carcinomas, urothelial and renal carcinomas, small cell bronchial carcinomas and squamous cell carcinomas of the skin [depending on the current drug approval]) which will be treated with ICI (PD-1/PD-L1) and potential radiation of metastases at Department of Radiation Oncology of Universitätsklinikum Erlangen.
  Interventions: Other: Conventional Therapy acc. to prevailing clincal approved schemes

INTERVENTIONS:
Other: Conventional Therapy acc. to prevailing clincal approved schemes — The study is observational. The treatment-plan of the underlying disease remains unchanged. The treatment of the patient is according to the prevailing clinical approved schemes at the respective entities. Blood will be drawn from patients at several time points during and after RT and ICI for detailed immunomonitoring of the patients.

SUMMARY:
Inhibitors of the programmed cell death protein 1 (PD-1)/PD-L1 immune checkpoint signaling pathway are already approved in the treatment of various tumor entities in relapsed or metastatic stages. Different exploratory trials suggest that the combination of radiotherapy and PD-1/PD-L1 inhibitors is highly effective, especially in oligometastatic stages and if all lesions are treated with ablative radiotherapy. In addition, the role of predictive biomarkers is becoming increasingly important for future therapy algorithms. First data, also from our group, indicate clearly that dynamic changes of immune cells and their activation markers in the peripheral blood (immune matrix) can be used as predictive biomarkers. During the planned STICI-02 trial predictive immune matrix derived from the STICI01 trial (NCT03453892) will be validated in the groups of patient suffering from HNSCC (palliative), NSCLC (separately palliative and adjuvant) and "other solid tumors" (including in particular esophageal carcinomas, urothelial and renal carcinomas, small cell bronchial carcinomas and squamous cell carcinomas of the skin [depending on the current drug approval]). Within the framework of scientific accompanying projects, the predictive value of markers in tumor tissue and of pattern radiomics analyses will be analyzed accompanying the immunophenotyping in peripheral blood. The side effects

ELIGIBILITY:
Inclusion Criteria:

* Patients treatable for HNSCC (palliative), NSCLC (separately palliative and adjuvant) or "other solid tumour"
* Indication for system therapy with a PD-1/PD-L1 inhibitor according to clinical standards
* Patients without or with radiation of one or more metastases
* Age at least 18 years

Exclusion Criteria:

* Melanoma patients
* Fertile patients who refuse effective contraception during study treatment
* Persistent drug and/or alcohol abuse
* Patients not able or willing to behave according to study protocol
* Patients in care
* Patients that are not able to speak German
* Patients which are imprisoned according to legal or governmental order

Both gender are included into the study, a maximum age was not defined.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study cohort consist of patients suffering from HNSCC (palliative), NSCLC (separately palliative and adjuvant) and "other solid tumors" (including in particular esophageal carcinomas, urothelial and renal carcinomas, small cell bronchial carcinomas and squamous cell carcinomas of the skin [depending on the current drug approval]) which will be treated with ICI (PD-1/PD-L1) and potential radiation of metastases at Department of Radiation Oncology of Universitätsklinikum Erlangen.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-04-30 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Overallsurvival | From inclusion till death of subject or up to 5 years, whichever came first.
  Prospective investigation of the survival of the patients.
Longitudinal Immunophenotype | Day 0 till progression or end of study up to 5 years or till change to conventional treatment without ICI, whichever came first.
  Longitudonal Immunophenotyping of the patients: Detection of about 30 distinct immune cell (sub)types together with their activation markers during treatement.
Predictors in pattern recognition analyses | Day 0 till progression or end of study up to 5 years or till change to conventional treatment without ICI, whichever came first.
  Identification of possible predictors in pattern recognition analyses from clinical imaging data sets.
Immune-associated side effects | Day 0 till progression or end of study up to 5 years or till change to conventional treatment without ICI, whichever came first.
  Detection of immune-associated side effects

SECONDARY OUTCOMES:
Detection of adverse events according to NCI CTAE (v4.0) | From date of inclusion to the trial until the date of first documented iRECIST progression or date of death from any cause, or till change to conventional treatment , whichever came first, assessed up to 5 years.
  The adverse effects of Immunecheckpoint and Radiotherapy is recorded by official questionaire
Progression free survival | From date of inclusion to the trial until the date of first documented iRECIST progression or date of death from any cause, whichever came first, assessed up to 5 yeras
  survival of the patient without progression of malignant disesase
Treatment response (according to RECIST and iRECIST criteria) | From date of inclusion to the trial until the date of first documented iRECIST progression or date of death from any cause, whichever came first, assessed up to 5 years
  RECIST and iRECIST criteria will used to analyse the response of the patient to the respective treatement
Attempt to establish an immune matrix of responding/non-responding patients | The analyses are conducted at time points before (day 0) and before every prescription of ICI (every 14 to 21 days) till progression or end of study up to 5 years or till change to conventional treatment without ICI.
  Analysis of clincal, MRI and imunnologic, molecular data to develop an biomarkermatrix with processes of machine learning

CONTACTS AND LOCATIONS:
Overall Officials: Markus Hecht, PD Dr., Study Director — Universitätsklinikum Erlangen, Department of Radiation Oncology; Udo S Gaipl, Prof. Dr., Principal Investigator — Universitätsklinikum Erlangen, Department of Radiation Oncology; Rainer Fietkau, Prof. Dr., Study Chair — Universitätsklinikum Erlangen, Department of Radiation Oncology; Benjamin Frey, PD Dr. Dr., Principal Investigator — Universitätsklinikum Erlangen, Department of Radiation Oncology
Locations (1):
- Department of Radiation Oncology, Universitätsklinikum Erlangen, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided